CLINICAL TRIAL: NCT03096015
Title: Intensive Interdisciplinary Treatment Program for Individuals With Stroke-Induced Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Elizabeth Hoover, Clinical Associate Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3174E
Record Dates: First submitted 2017-03-21; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Within-subjects Group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive Treatment for Aphasia (Experimental)
  Interventions: Behavioral: Intensive Comprehensive Aphasia Program

INTERVENTIONS:
Behavioral: Intensive Comprehensive Aphasia Program

SUMMARY:
An intensive, interdisciplinary treatment program was administered during the summer as part of regular clinic services in the Aphasia Resource Center (ARC) at Sargent College. This program was run program as described for three years. Not more than six native English speakers with mild or moderate profiles of aphasia and multidisciplinary rehabilitation needs (OT,PT, SLP and nutrition) were recruited from the Boston community to participate in an intensive interdisciplinary treatment program for four weeks during the month of June 2013. The program consists of approximately six hours of interdisciplinary treatment each day, five days per week over a four-week interval. Treatment is individualized using current evidence-based treatment approaches, which are commonly accepted protocols in clinical practice and will be administered by clinical faculty and staff from Speech-Language and Hearing Sciences, Occupational Therapy (OT), Physical Therapy (PT), the Center for Neurorehabilitation and Nutrition. Segments of these types of treatments are available for a small fee as part of our service in the Aphasia Resource Center; however, this comprehensive, interdisciplinary program is not available of this research study.

Approximately 30 hours of therapy per week are provided -- 6 hours per day over 5 days consisting of Speech-language Pathology, Physical Therapy, Occupational Therapy, and Nutrition Counseling.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild or moderate profile of aphasia secondary to a single stroke, as diagnosed by a certified speech-language pathologist.
* Must be able to demonstrate auditory comprehension at a level that is functional for conversation.
* Must demonstrate mobility or sensory deficits as a result of the stroke.
* Must demonstrate cardiac/nutritional needs.
* Must be able to ambulate without the physical assistance of another person for at least 500 feet.
* Must be able to negotiate elevator and stairs independently
* Must be able to manage bathroom needs without assistance.
* Must be more than twelve months post-onset of stroke.
* Must be between 18 and 75 years of age.
* Must be native speakers of English
* Must have 8th grade level of education or higher.
* Must have adequate vision for functional reading
* Must have adequate hearing for conversation

Exclusion Criteria:

* Subjects who meet the above inclusion criteria, but who are also bilingual, and/or have concomitant neurological disease will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale (to assess change) | 1 month pre intervention, immediately prior to intervention, the week post intervention, 3 months after intervention was completed
  QoL indicator for stroke survivors
Canadian Occupational Performance Measure (to assess change) | 1 month pre intervention, immediately prior to intervention, the week post intervention, 3 months after intervention was completed
  Measures participation and satisfaction in meaningful activities

SECONDARY OUTCOMES:
Goal Attainment Scaling (to assess change) | 1 month pre intervention, immediately prior to intervention, the week post intervention, 3 months after intervention was completed
  Measures attainment of individualized/personal community-based goals

IPD SHARING:
Plan to Share IPD: No